CLINICAL TRIAL: NCT04299087
Title: Changes in Cortical Oscillations Induced by Repetitive Transcranial Magnetic Stimulation (rTMS) Therapy in Patient Populations With Tremor
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for Dystonia and Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201902838; R01NS058487 (NIH)
Record Dates: First submitted 2020-02-28; First posted 2020-03-06 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Dystonia; Tremor
MeSH Terms: conditions — Dystonia; Tremor | interventions — Transcranial Magnetic Stimulation; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Dystonia and/or tremor (Experimental): Adults with a diagnosis of dystonia and/or tremor
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)
- Control (Experimental): Healthy adults without a history of any neurological disorder, with a similar age distribution and sex ratio as the dystonia and/or tremor group
  Interventions: Other: Control group

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation (rTMS) — Repetitive transcranial magnetic stimulation (rTMS) is a form of brain stimulation therapy using a magnet to target and stimulate certain areas of the brain.
  Arms: Dystonia and/or tremor
Other: Control group — No application of rTMS
  Arms: Control

SUMMARY:
The study will include subjects diagnosed with Dystonic Tremor (DT), Essential Tremor (ET), and healthy controls in the age range of 21-80 years. Electroencephalography (EEG) will be used as the primary outcome measure. Transcranial Magnetic Stimulation (TMS) will be used over the motor cortices or cerebellar cortices as an intervention that is expected to have short-term (less than an hour) electrophysiological effects.

DETAILED DESCRIPTION:
The primary goal of this study is to compare differences in cortical activity of patients with tremor before and after applying a session of rTMS. Specifically, the investigators will apply rTMS to the primary motor cortex (M1) as our group and others have shown abnormal function of the region. Moreover, a study shows that targeting of M1 and the dorsal premotor cortex (dPMC) with rTMS results in a trend towards improved clinical outcome in patients with focal hand dystonia and cervical dystonia. The central hypothesis of this study is that rTMS can modify cortical oscillations in patient populations with tremor and that the investigators will be able to detect these changes with the use of Electroencephalography (EEG). By applying inhibitory rTMS to the motor cortices, the investigators may expect a shift in cortical oscillations towards normal activity.

ELIGIBILITY:
Inclusion Criteria for Dystonia and/or tremor:

- Diagnosis of Dystonia and/or tremor according to the Consensus Statement of the Movement Disorders Society

Exclusion Criteria Dystonia and/or tremor:

* Pregnancy
* Active seizure disorder
* Presence of a metallic object such as a pacemaker, implants, metal rods, and hearing aid
* History of stroke

Inclusion Criteria for Healthy controls

- There is no history of any neurological disorders.

Exclusion Criteria for Healthy controls

* Pregnancy
* Any neurological disorders
* Presence of a metallic body in their brain
* History of stroke

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Vaillancourt, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dystonia and/or Tremor | Control
Started | 11 | 1
Completed | 9 | 0
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dystonia and/or Tremor | Control | Total
Number analyzed (Participants) | 11 | 1 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 7 | 0 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.583 (11.172) | 66 (0) | 63.583 (11.172)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 8
  Male | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 1 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Assessment Using MoCA Version 7.1 Scores
Description: Montreal Cognitive Assessment Version 7.1 was used to assess cognitive ability. This scales is score from a range of 0 to 30 with a score of 24 or less indicating mild cognitive impairment. Moderate cognitive impairment is indicated by a score of 18-23 and severe impairment is a score of 10 or less. Overall, a higher number indicates better cognitive ability.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dystonia and/or Tremor | Control
Number analyzed (Participants) | 11 | 1
units on a scale | 25.45 (3.78) | 27 (0)

ADVERSE EVENTS:
Time Frame: approximately 7 days a part
Arm/Group | Dystonia and/or Tremor | Control
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/1
Other Adverse Events (participants affected / at risk) | 0/11 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/87/NCT04299087/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/87/NCT04299087/ICF_001.pdf